CLINICAL TRIAL: NCT04314856
Title: Sigma-1 Receptors: A Novel Clinical Target in Fragile X Syndrome
Brief Title: Novel Clinical Target in Fragile X Syndrome
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal investigator left institution
Sponsor: Guido A. Davidzon, MD, SM (Other)
Responsible Party: Sponsor-Investigator, Guido A. Davidzon, MD, SM, Associate Professor of Radiology/Nuclear Medicine & Molecular Imaging, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB 50016
Record Dates: First submitted 2020-03-11; First posted 2020-03-19 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Fragile X Syndrome (FXS)
Keywords: FXS
MeSH Terms: conditions — Fragile X Syndrome | interventions — 6-(3-fluoropropyl)-3-(2-(azepan-1-yl)ethyl)benzo(d)thiazol-2(3H)-one

STUDY DESIGN:
Intervention Model Description: 15 male subjects with FXS will be compared to 5 healthy volunteers who will be the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fragile X Syndrome (Experimental): Adult males aged 18-30 years diagnosed with FXS will undergo a PET/MRI scan using 18F-FTC-146 to determine sigma-1 receptor density.
  These participants will only be administered once with 18F-FTC-146.
  Interventions: Drug: 18F-FTC-146
- Healthy Volunteers (Control) (Experimental): Adults aged 18-65 years undergo a PET/MRI scan using 18F-FTC-146 to determine sigma-1 receptor density.
  Test-retest studies will be performed where these individuals will each be injected twice with 18F-FTC-146.
  Interventions: Drug: 18F-FTC-146

INTERVENTIONS:
Drug: 18F-FTC-146 — 18F-FTC-146 is a PET radiopharmaceutical that can be used to determine sigma-1 receptor density.
  Other Names: FTC146

SUMMARY:
Fragile X syndrome (FXS) is the most common genetic cause of autism spectrum disorder (ASD). The investigators wish to examine brain distribution of sigma-1 receptors in young adult males with FXS using 18F-FTC-146 PET. This project will study the distribution of sigma-1 receptors in 15 young (18-30 years) male adults with FXS compared to 5 healthy adult volunteers.

DETAILED DESCRIPTION:
In this study, we measured sigma-1 receptor density in the regions of interest in brain known to be involved in executive functioning and cognition using 18F-FTC-146 PET. We then compared S1R density in areas ROIs not involved in executive functioning and cognition. This provided a framework for predicting functional impairment based on brain-behavior relationships.

The study had two aims. The first aim was to evaluate the reliability of 18F-FTC-146 brain uptake in healthy controls under test and retest conditions to establish a baseline measure of S1R density and quantify regional brain uptake of radiotracer in five healthy adults. The second aim was to characterize S1R density in brains of young adult males with FXS which will then be compared to healthy volunteers.

This was the very first PET study to image sigma-1 receptor density in participants with fragile X syndrome, thereby testing whether altered receptor density is present in brain in fragile X syndrome patients when compared to healthy volunteers. If confirmed, the current study would have provided compelling clinical-translational support for an important pathophysiological mechanism of cognition and executive function. The study had considerable potential for advancing the neurobiological understanding of fragile X syndrome in humans.

ELIGIBILITY:
INCLUSION CRITERIA

Inclusion criteria for healthy volunteers:

1. Ages 18-65
2. Either gender and all ethno-racial categories
3. Capacity to provide informed consent
4. Female participants are expected to use an effective method of birth control throughout the study which includes: hormonal methods (birth control pills, patches, injections, vaginal ring or implants), barrier method (condom or diaphragm) used with spermicide, intrauterine device (IUD), or abstinence (no sex)
5. Can travel to Stanford for 2 scan days.

Inclusion criteria for individuals with FXS:

1. Males who are physically healthy
2. Aged between 18 and 30 years inclusive
3. Can travel to Stanford for a 2-day visit.
4. IQ between 40 and 80 points.
5. Ability to remain seated for more than 10 minutes.
6. Have an established genetic diagnosis of FXS (full mutation with evidence of aberrant methylation of the FMR1 gene, confirmed by genetic testing).

EXCLUSION CRITERIA

Exclusion criteria for healthy volunteers:

1. Any current or lifetime psychiatric diagnosis
2. Current or past use of psychotropic medication for purposes of treating a mental illness
3. Pregnant or nursing females
4. Major medical or neurological problem, including anemia (Hb , 12 g/dl in women and <14 g/dl in men) (e.g., unstable hypertension, seizure disorder, head trauma)
5. Current diagnosis of vasculopathy or Raynouds
6. Participant is unable to tolerate being off of anticoagulant medication during study
7. Positive urine screen for illicit drugs
8. Presence of metal in the body that is contraindicated for MRI scans
9. Current exposure to radiation in the workplace, or history of participation in nuclear medicine procedures does not exceed defined annual limits
10. Stanford University student status (i.e., we will exclude students such as undergrads, grad students and postdocs that currently attend at Stanford University)

Exclusion criteria for individuals with FXS:

1. Any contraindication for MRI scanning procedures (metal in body, braces, claustrophobia, etc.)
2. No history of with substance abuse, traumatic brain injury and
3. BMI greater than 18.5
4. Diagnosis of a known genetic disorder (other than FXS).
5. Active medical problems such as unstable seizures, congenital heart disease, endocrine disorders.
6. Significant sensory impairments such as blindness or deafness.
7. DSM-5 diagnosis of other severe psychiatric disorder such as bipolar disorder or schizophrenia.
8. Pre-term birth (<34 weeks' gestation) or low birth weight (<2000g).
9. Current use of benzodiazepines. Individuals who are taking concomitant psychoactive medications will be tracked and examined in post-hoc analyses, given that it is extremely difficult to recruit individuals who are medication-free or who are willing to go off those medications prior to entering the study.
10. Current exposure to radiation in the workplace, or history of participation in nuclear medicine procedures does not exceed defined annual limits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For FXS only: Participants must be male adults between 18 and 30 years with Fragile X-syndrome
Enrollment: 0 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of concordant readings of regional brain uptake of radiotracer [18F]FTC-146 as a measure of reliability under test-retest conditions | Up to 6 hours per scan performed on Day 0 (Test) and Day 7 (Retest)
  Regional brain uptake of [18F]FTC-146 will be analyzed by kinetic modeling with metabolite-corrected arterial input functions to establish stability and reproducibility of [18F] FTC-146 in humans under test and retest conditions.
  This outcome will be assessed in healthy volunteers only.
Difference in Non-displaceable Binding Potential (BPND) of [18F]FTC-146 in fragile X syndrome (FXS) patients relative to healthy volunteers | Up to 6 hours per scan performed on Day 0 (both groups) and Day 7 (healthy volunteers)
  Binding potential provides an estimate of the S1R receptor distribution and affinity of [18F]FTC-146 to the S1R receptors. Binding potential measurements will be compared between participants with fragile X syndrome and control group with healthy volunteers to assess if there is a difference. Binding Potential (BPND) is estimated as the distribution volume ratio (DVR) -1.
  DVR's of tracers are used in PET receptor studies where the radiopharmaceutical can be specifically bound to receptors; nonspecifically bound to other macromolecular components, or free in tissue (FT). DVR is calculated using a Logan Plot, which uses the dynamic PET images obtained during imaging and compartment modeling to graphically analyze by linear regression pharmacokinetic data for radiopharmaceuticals that undergo 'reversible' uptake.
  Healthy volunteers will have scans at Day 0 and Day 7, and FXS patients will have a single scan on day 0. All scans will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Davidzon, MD SM, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cipriano PW, Lee SW, Yoon D, Shen B, Tawfik VL, Curtin CM, Dragoo JL, James ML, McCurdy CR, Chin FT, Biswal S. Successful treatment of chronic knee pain following localization by a sigma-1 receptor radioligand and PET/MRI: a case report. J Pain Res. 2018 Oct 12;11:2353-2357. doi: 10.2147/JPR.S167839. eCollection 2018. PMID 30349360
- [Background] Shen B, Park JH, Hjornevik T, Cipriano PW, Yoon D, Gulaka PK, Holly D, Behera D, Avery BA, Gambhir SS, McCurdy CR, Biswal S, Chin FT. Radiosynthesis and First-In-Human PET/MRI Evaluation with Clinical-Grade [18F]FTC-146. Mol Imaging Biol. 2017 Oct;19(5):779-786. doi: 10.1007/s11307-017-1064-z. PMID 28280965
- [Background] Hjornevik T, Cipriano PW, Shen B, Park JH, Gulaka P, Holley D, Gandhi H, Yoon D, Mittra ES, Zaharchuk G, Gambhir SS, McCurdy CR, Chin FT, Biswal S. Biodistribution and Radiation Dosimetry of 18F-FTC-146 in Humans. J Nucl Med. 2017 Dec;58(12):2004-2009. doi: 10.2967/jnumed.117.192641. Epub 2017 Jun 1. PMID 28572487